CLINICAL TRIAL: NCT03927027
Title: ARM: Axillary Reverse Mapping - A Prospective Trial to Study Rates of Lymphedema and Regional Recurrence After Sentinel Lymph Node Biopsy and Sentinel Lymph Node Biopsy Followed by Axillary Lymph Node Dissection With and Without Axillary Reverse Mapping
Brief Title: Axillary Reverse Mapping in Preventing Lymphedema in Patients With Breast Cancer Undergoing Axillary Lymph Node Dissection
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A221702; NCI-2018-02445 (Registry Identifier: NCI Clinical Trial Reporting Program); UG1CA189823 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Neoplasms | interventions — iso-sulfan blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (ALND) (Active Comparator): Patients receive isosulfan blue SC and undergo ALND.
  Interventions: Drug: Isosulfan Blue; Procedure: Axillary Lymph Node Dissection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (ARM, ALND) (Experimental): Patients undergo ARM. Patients then receive isosulfan blue and undergo ALND as in Group I.
  Interventions: Drug: Isosulfan Blue; Procedure: Axillary Lymph Node Dissection; Procedure: Mapping; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Isosulfan Blue — Given SC
Procedure: Axillary Lymph Node Dissection — Undergo ALND
  Other Names: ALND; axillary dissection
Procedure: Mapping — Undergo ARM
  Arms: Group II (ARM, ALND)
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well axillary reverse mapping works in preventing lymphedema in patients with breast cancer undergoing axillary lymph node dissection. Axillary reverse mapping may help to preserve the lymph node drainage system around the breast so as to prevent lymphedema after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the occurrence of post-surgery lymphedema by conical geometric measures in clinical T1-3, N0-3, M0 breast cancer patients undergoing axillary surgery and randomized to Group 1 (no axillary reverse mapping [ARM]) versus Group II (ARM).

SECONDARY OBJECTIVES:

I. To compare between the study groups the lymphedema symptom intensity and distress as measured by the Lymphedema Symptom Intensity and Distress Survey-Arm (LSIDS-A).

II. To evaluate the technical success of performance of ARM procedure: Identification of ARM lymphatics, and the ability to spare or reapproximate ARM lymphatics.

III. To compare the rate of regional recurrence between patients randomized to receive ARM versus no ARM.

EXPLORATORY OBJECTIVES:

I. To assess the occurrence of lymphedema as a function of radiotherapy use and targets.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive isosulfan blue subcutaneously (SC) and undergo axillary lymph node dissection (ALND).

GROUP II: Patients undergo ARM. Patients then receive isosulfan blue and undergo ALND as in Group I.

After completion of study, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of Disease: cT1-3 patients undergoing axillary surgery who additionally meet one of the following conditions:

  * Clinically node negative patients undergoing mastectomy and sentinel lymph node biopsy (SLNB) with possible axillary lymph node dissection (ALND) if SLNB is positive. If ALND is performed during a separate operation, ARM procedure must be repeated. Clinically node negative is defined by i) negative clinical exam and/or ii) negative axillary US and/or iii) negative needle biopsy of sonographically suspicious axillary nodes as applicable to each case.
  * Clinically node positive patients as determined by needle biopsy and planned for ALND regardless of type of breast surgery.
  * Patients will be staged according to the TNM staging system.
* Prior Treatment: No prior axillary surgery except needle biopsy or concurrent SLNB.

  o Prior neoadjuvant chemotherapy is allowed but must be completed at least 2 weeks before registration.
* No prior history of ipsilateral breast cancer (invasive or ductal breast carcinoma in situ [DCIS]). Lobular breast carcinoma in situ (LCIS) and benign disease are allowed. (May have neoadjuvant chemotherapy which must be completed 2 weeks before registration).
* No bilateral invasive breast cancer.
* No matted nodes.
* No history of lymphedema of either arm.
* No known allergies blue dyes, including make-up containing blue dye.
* In order to complete the mandatory patient-completed measures, participants must be able to speak and/or read English.
* Female :

Men are excluded from this study because the number of men with breast cancer is insufficient to provide a statistical basis for assessment of effects in this subpopulation of people with breast cancer.

* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
* Creatinine: =< 1.5 x upper limit of normal (ULN).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of upper extremity (UE) lymphedema | Up to 36 months post surgery
  Will be assessed by the Lymphedema Symptom Intensity and Distress Survey-Arm (LSIDS-A). The LSIDS-A questionnaire contains two different scales for intensity and distress measured from 1 (slight) to 5 (severe). The LSIDS-A questionnaire scores for swelling in the arm, decreased physical activity, pain in the arm, and loss of confidence in one's body will be evaluated for the change of baseline to 36 months using a two-sample, two-sided t-test.

SECONDARY OUTCOMES:
Change in health-related quality of life: LSIDS-A questionnaire scores | Baseline to 36 months
  Will be assessed by the Lymphedema Symptom Intensity and Distress Survey-Arm (LSIDS-A). The LSIDS-A questionnaire scores at each time point, as well as the change from baseline will be compared between groups by a two-sample, two-sided t-test. If there is evidence of non-normality (via Shapiro-Wilk testing), will use a non-parametric procedure such as Wilcoxon rank sum test. Further analysis will include linear mixed model using data from all time points to compare the LSIDS-A questionnaire scores between the two treatment groups over time adjusting for other baseline characteristics. Will evaluate the pattern of missing data. If the drop-out rate is higher than expected, methods proposed by Hogan and Laird will be used to assess whether the presence of drop-outs affects inferences obtained from the repeated measures analyses. Appropriate methods will be used to address missingness.
Incidence of regional recurrence | Up to 3 years
  The technical success will be summarized using a binomial point estimate and 95% confidence interval (CI) and will be compared using a two-sample test of proportions.
Technical success of performance of axillary reverse mapping (ARM) procedure (defined as identification of ARM lymphatics, and the ability to spare or reapproximate ARM lymphatics) | Up to 3 years
  The cumulative incidence of regional recurrence will be summarized using the cumulative incidence function treating death without regional recurrence as the competing risk. Similar analysis methods described for the primary endpoint will be used to compare the cumulative incidence of regional recurrence between group I and II.

CONTACTS AND LOCATIONS:
Overall Officials: V. Suzanne Klimberg, MD, PhD, Study Chair — University of Texas
Locations (96):
- United States (96):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Shaw Cancer Center, Edwards, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Anne Arundel Medical Center, Annapolis, Maryland
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Cancer Institute at Saint Francis Hospital, East Hills, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Pluta Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Geisinger South Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - UTMB Health Angleton Danbury Campus, Angleton, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levy AS, Murphy AI, Ishtihar S, Peysakhovich A, Taback B, Grant RT, Ascherman JA, Feldman S, Rohde CH. Lymphatic Microsurgical Preventive Healing Approach for the Primary Prevention of Lymphedema: A 4-Year Follow-Up. Plast Reconstr Surg. 2023 Feb 1;151(2):413-420. doi: 10.1097/PRS.0000000000009857. Epub 2022 Nov 15. PMID 36696330